CLINICAL TRIAL: NCT06931197
Title: Why Wait? Initiating Contingency Management in Traumatically Injured Patients During Hospitalization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-2025-012
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Contingency Management; Methamphetamine Use Disorder
Keywords: Contingency management; Methamphetamine Use Disorder; Contingency management during acute hospitalization; Contingency management in Trauma Injured Patients

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the CM intervention group and for the total of 12 weeks, he/she will be followed up two times a week during the hospitalization and up to three times per week as an outpatient to engage in intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency management intervention (Experimental): Intervention is total of 12 weeks. During the hospitalization, participants will be visited by study personnel and will be asked to complete a urine drug screen that will screen for presence of methamphetamine on Mondays/Thursdays or Tuesdays/Fridays (M/Th or T/F). Once discharged, participants will be asked to come into the out patient clinic 2 times per week (M/Th or T/F) to complete a urine drug screen that will screen for presence of methamphetamine. If the specimen is negative for methamphetamine, the participants will be rewarded. Participants will also be asked to complete the Treatment Effectiveness Assessment (TEA) with study personnel.
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — If the urine sample is methamphetamine negative, participant will be positively reinforced and offered incentives. Participants immediately draw the reinforcement slip of paper to receive a prize from a selection kept on-site. Approximately 50% of the slips offer written praises (i.e. "great job!"). The other 50% of slips are the divided between low value (i.e. food gift cards, bus passes), medium value (i.e. prepaid cellphone, clothing gift cards), and a few large value rewards (i.e. electronic tablet, jewelry). Should the sample be positive for methamphetamine, no reinforcement and/or incentive to be provided. Participant will be encouraged to continue to participate in CM program and follow-up on the next CM date.

SUMMARY:
This clinical trial is to implement contingency management (CM) as an intervention tool to address methamphetamine use and will be initiated during inpatient acute hospitalization in trauma injured patients.

The goals are:

* Gather effectiveness data on a CM program for participants in Hawaii who use methamphetamine during hospitalization and following discharge due to trauma injury
* To assess participant perspectives on engaging with a CM program based at a Level 1 Trauma Center. Researches will assess both patient-reported and biologically-confirmed medium-term program effectiveness and conduct qualitative interviews with participants post-program.
* To assess the rate of leaving against medical advice (AMA) and treatment completion in acute hospital setting in participants.
* To assess the optimal timing of CM initiation for traumatically injured hospitalized patients by comparing patient outcomes (i.e. duration of CM participation and rates of CM program completion and providing negative urine samples) to NCT06532370 where CM was initiated after discharge from the hospital.

For total of 12 weeks, participants will:

* Be visited on Mondays/Thursdays or Tuesdays/Fridays by the research team to complete urine analysis during the hospitalization
* Visit a follow up clinic up to 2 times per week on Mondays/Thursdays or Tuesdays/Fridays to complete urinalysis following discharge from the hospital
* Complete Treatment Effectiveness Assessments at 6 and 12 weeks
* Engage in qualitative interview at the end of the CM program

ELIGIBILITY:
Inclusion Criteria:

* Admitted trauma patients
* Age greater than 18 years old
* Urine drug screen positive for methamphetamines during the current hospitalization
* Report at least weekly methamphetamine use
* First methamphetamine use greater than 6 months prior to injury
* Report at least 4 Diagnostic and Statistical Manual of Mental Disorders 5th Edition, Amphetamine-Type Substance Use Disorder symptoms (at least moderate disease)
* Glasgow Coma Scale ≥13 upon arrival to the emergency department
* Ability to understand and participate in study procedures
* Ability to communicate in English
* Expected discharge date within 45 days on the day of screening / recruitment

Exclusion Criteria:

* Active psychosis (reporting auditory or visual hallucinations)
* Under ongoing cardiorespiratory monitoring
* Evidence of moderate or severe traumatic brain injury
* Patients who are known to be pregnant
* Prisoners
* Individuals incarcerated at the time of their hospitalization
* Individuals lacking capacity to provide, or are otherwise unable or unwilling to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Effectiveness Assessments (TEA) at 6- and 12-weeks post-enrollment | From enrollment to 6 and 12 weeks
  TEA (Treatment Effectiveness Assessment) at 6- and 12-weeks post-enrollment to assess both patient-reported medium-term program effectiveness. TEA asks individuals to respond to changes in four domains following a drug treatment program: Substance use, health, lifestyle, and community. The score for each domain can range from 1 (no change or not much) to 10 (much better), for total score of 4-40. This score allows for the prioritization of each participants values, and therefore does not require strict abstinence to demonstrate benefit from drug treatment.

SECONDARY OUTCOMES:
Conduct qualitative interviews with participants post-program | At the end of the treatment at 12 weeks
  Interviews will be conducted as semi-structured qualitative interviews with participants post-program and will be transcribed and analyzed using a Template Analysis approach. Coders will conduct coding of the interview data to ultimately identify themes that will be used as the basis for interpretation. The final analysis of the qualitative data will include contrasts and comparisons made across interviews to examine overlaps and divergences across any relevant sub-samples (i.e. sex, age). Results will present thematic patterns, how frequently each code occurs, and any contradictory evidence. This will allow for the identification of common themes and perspectives, which will provide necessary cultural insights and possible adaptations for further implementation efforts.

OTHER OUTCOMES:
Assessment of rate of AMA and treatment completion in acute hospital setting in participants | From enrollment to the end of treatment at 12 weeks
  To assess the rate of AMA and treatment completion in acute hospital setting in participants
  To assess the optimal timing of CM initiation for trauma injury hospitalized patients by comparing patient outcomes to the Schumann's pilot project 2024 (7/2024-6/2025) (NCT06532370 - Implementing a Contingency Management Program Addressing Methamphetamine Use For and With the People of Hawaii). We will compare the duration of CM participation and the rates of CM program completion and providing negative urine samples.

CONTACTS AND LOCATIONS:
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No